CLINICAL TRIAL: NCT00353054
Title: A Double-Blind, Randomized, Placebo Controlled, Parallel Group Study to Evaluate the Effect of Calcium/Vitamin D Supplementation (Caltrate 600+ D) on Body Weight and Fat Loss in Overweight and Obese Individuals on a Weight-Reducing Program.
Brief Title: Effect of Calcium/Vitamin D Supplementation on Body Weight and Fat Loss.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-02-01
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2006-07-17 (Estimated); Status verified 2002-11

CONDITIONS: Obesity; Overweight
Keywords: Caltrate; Lipoproteins; Glucose; Insulin; Blood pressure; Body fat; Body weight; Women; Diet; Macronutrients
MeSH Terms: conditions — Obesity; Overweight; Insulin Resistance; Body Weight | interventions — Fumigant 93

INTERVENTIONS:
Drug: Caltrate® 600 + D
Behavioral: Weight loss intervention

SUMMARY:
The aim of this study was to assess the effect of calcium/vitamin D supplementation (Caltrate 600 +D®) on body weight loss during a weight-reducing program

DETAILED DESCRIPTION:
The effect of a calcium supplementation on body weight loss is inconclusive and some studies have suggested that adequate calcium intake can have a favourable effect on some metabolic variables. The objectives of this study were to evaluate the impact of (Caltrate 600 + D ®) on body composition and various indicators of metabolic health in overweight and obese females characterised by a usual low daily calcium intake, on a weight-reducing program.

The main hypotheses of this study were:

* Caltrate 600 +D® increases body weight and fat mass losses of individuals on a weight-reducing program.
* Caltrate 600 +D® improves the metabolic profile of these subjects, independently of variations promoted by body fat loss.

ELIGIBILITY:
Inclusion Criteria:

* Daily calcium intake below 800mg/day
* Stable body weight
* Body mass index (BMI) between 27-40kg/m2
* Less than 3 periods of 20 minutes of physical exercise/week
* General good health
* Normal blood pressure values
* Normal cholesterol levels
* Normal thyroid hormone levels
* No participation in another clinical trial within 6 months of screening
* Coffee consumption ≤ 5 cups/day.

Exclusion Criteria:

* Breast feeding, pregnant or menopaused women
* Use of calcium supplements within 30 days of screening
* Cholesterol levels requiring pharmaceutical treatment
* Smoking
* Use of medication that could affect body weight

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80
Dates: Start 2003-01; Study Completion 2005-07

PRIMARY OUTCOMES:
Body weight and fat mass loss at the end of the 15-week weight loss supplemented intervention.

SECONDARY OUTCOMES:
Change in metabolic variables at the end of the 15-week calcium/vitamin D supplemented weight loss intervention
Change in energy/macronutrient intake at the end of the 15-week calcium/vitamin D supplemented weight loss intervention

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Tremblay, PhD, Principal Investigator — Laval University
Locations (1):
- Université Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Major GC, Alarie FP, Dore J, Tremblay A. Calcium plus vitamin D supplementation and fat mass loss in female very low-calcium consumers: potential link with a calcium-specific appetite control. Br J Nutr. 2009 Mar;101(5):659-63. doi: 10.1017/s0007114508030808. PMID 19263591